CLINICAL TRIAL: NCT04503109
Title: Spinal Cord Stimulation in the Treatment of Chronic, Intractable Pain Using the Nalu™ Neurostimulation System
Acronym: nPower™-US
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nalu Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAL-01-2020-US
Record Dates: First submitted 2020-08-03; First posted 2020-08-07 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Pain, Chronic; Pain, Intractable; Pain, Back
Keywords: Spinal Cord Stimulation; Chronic Leg and Back Pain; Failed Back Surgery Syndrome (FBSS)
MeSH Terms: conditions — Chronic Pain; Pain, Intractable; Back Pain; Failed Back Surgery Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Nalu SCS System (Other): All eligible subjects will receive the Nalu Neurostimulation System
  Interventions: Device: Nalu Neurostimulation System

INTERVENTIONS:
Device: Nalu Neurostimulation System — The Nalu Neurostimulation System is a Spinal Cord Stimulation system

SUMMARY:
The Nalu Neurostimulation System is capable of delivering multiple therapy options to address patient needs. The study will confirm the efficacy, safety, comfort and compliance with the Nalu Neurostimulation System in adult subjects with chronic pain in the legs and back. Patients who have been diagnosed with failed back surgery syndrome (FBSS) and meet other study eligibility criteria will be enrolled in the study to receive the Nalu Neurostimulation System.

DETAILED DESCRIPTION:
The study is a prospective, multi-center, open-label, single-arm clinical study with each subject serving as their own control. The study will confirm device efficacy, safety, comfort and compliance with the system.

Subjects who meet the protocol specified eligibility criteria and provide documented informed consent will be considered for study participation. There are three phases in the study: Screening/Baseline Phase, Trial Phase, Permanent Implant Phase. On confirmation of eligibility during the screening/baseline phase, subjects will enter the Trial Phase where they will undergo a trial with the Nalu Neurostimulation System. Trials will be done per standard clinical practice and per system IFU. Subjects receiving at least 50% reduction in their back pain, during the trial phase, will continue to the permanent implant phase.

Eligible subjects will receive the Nalu Neurostimulation System per standard surgical and medical practices and will be programmed for stimulation with one or more therapies to optimize pain reduction. All subjects receiving a permanent implant will be followed for 3-months post device activation. They will visit the clinic at 1 month and 3-months follow-up and programming, as required. Adverse Event data will also be collected to support a safety endpoint.

Multiple outcome domains will be captured throughout the study to confirm system performance and subject response to the device. These include Visual Analogue Scale (VAS) for pain, Numeric Rating Scales for pain, EQ-5D (QoL), the Oswestry Disability Index (ODI), PROMIS Sleep Disturbance SF, Beck's Depression Index (BDI), pain and paresthesia maps, pain and wearability diaries.

At study completion, subjects will return to standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 21 and 80 years of age at enrollment.
2. Subject has chronic (defined as at least 6 months duration), intractable neuropathic pain of legs and/or back; any nociceptive pain must be less prominent than the neuropathic pain.
3. Subject's pain is unresponsive to conservative treatment options.
4. Subject has a VAS Score of at least 6 in the back and/or leg at screening.

Exclusion Criteria:

1. Subject currently has an active implantable medical device such as a drug pump, spinal cord stimulator, sacral nerve stimulator, deep brain stimulator, and/or cardiac pacemaker.
2. Subject has previously failed SCS therapy (either trial system evaluation or permanent implant).
3. Subject has had an ablative procedure directed at the spinal cord including the dorsal root entry zone (DREZ) or dorsal root ganglion (DRG).
4. Subject has pain in another anatomic region besides the leg(s) and back that would interfere with their ability to accurately report pain (e.g. hip joint pain).
5. Subject has a medical condition that would prevent them from participating in the current study per investigator's or medical monitor's judgment.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Responders at 3-months | 3 months
  Number of subjects who have 50% or greater pain reduction from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Martin, Study Director — Nalu Medical
Locations (8):
- United States (8):
  - CA Ortho and Spine, Larkspur, California
  - IPM Medical Group, Inc., Walnut Creek, California
  - International Spine, Pain and Performance Center, Washington D.C., District of Columbia
  - The Orthopaedic Institute, Gainesville, Florida
  - Southwest Florida Pain Center, Port Charlotte, Florida
  - Alliance Spine and Pain, Atlanta, Georgia
  - Neuroscience Research Center, Overland Park, Kansas
  - SSM Health, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No